CLINICAL TRIAL: NCT00137813
Title: Phase II Study of Bevacizumab and Docetaxel (AvaTax) in Metastatic Esophagogastric Cancer
Brief Title: Avastin and Taxotere for Esophagogastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-179
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Bevacizumab; Docetaxel; AvaTax; Metastatic Esophagogastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Docetaxel; Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — Given intravenously once a week for 3 out of four weeks for a minimum of 8 weeks and maximum of a year and a half
  Other Names: AvaTax
Drug: Bevacizumab — Given intravenously once a week for every other week for a minimum of 8 weeks and a maximum of a year and a half

SUMMARY:
The purpose of this study is to determine what effects (good and bad) bevacizumab (Avastin) and docetaxel (Taxotere), used in combination, have on metastatic gastric and esophageal cancer.

DETAILED DESCRIPTION:
Bevacizumab will be administered intravenously in an outpatient clinic once a week, every other week. Docetaxel will also be administered intravenously in the outpatient clinic once a week for three out of four weeks. Blood tests and vital signs will be performed weekly.

After the first eight weeks of therapy a CT scan will be performed to determine and assess the progress of the disease. If therapy is continued, radiological procedures will be performed at week 16 and every 8 weeks thereafter.

Treatment will be given for a minimum of 8 weeks, as long as the patient does not experience unacceptable side effects. Chemotherapy will continue for a year and a half as long as the cancer is responding and there are no unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable or metastatic stage IV esophageal or gastric carcinoma
* Measurable disease greater than or equal to 1cm by spiral computed tomography (CT) scan or greater than or equal to 2cm by other radiographic technique
* ECOG performance status 0-2
* One prior chemotherapy for metastatic disease permitted
* White blood cell count greater than or equal to 3,000/mm
* Absolute neutrophil count greater than or equal to 1,500/mm3
* Platelet count greater than or equal to 100,000/mm3
* Hemoglobin greater than or equal to 8.0g/dl
* Creatinine less than 2.0mg/dL
* Total bilirubin less than 1.9mg/dL

Exclusion Criteria:

* Pregnant or lactating women
* History or evidence of central nervous system (CNS) disease
* Other active malignancies other than non-melanoma skin cancer or in-situ cervical cancer
* History of severe hypersensitivity to docetaxel, bevacizumab or drugs formulated with polysorbate 80.
* Current, recent or planned treatment with standard chemotherapy, radiation therapy or another experimental therapy.
* History of other disease or metabolic dysfunction.
* Serious, non-healing wound, ulcer, or bone fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-08; Primary Completion 2006-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall response and safety of the combination docetaxel and bevacizumab in patients with esophageal or gastric cancer | 3 years

SECONDARY OUTCOMES:
To evaluate the duration of response, progression-free and overall survival of patients with esophageal or gastric cancer treated with docetaxel and bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Peter Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts